CLINICAL TRIAL: NCT02915133
Title: Correlation of Structural and Visual Function Changes in Myopia Foveoschisis Patients Undergoing Macular Buckle Surgery
Brief Title: The Relationship Between Structure and Visual Function in Myopia Foveoschisis
Status: Suspended | Type: Observational
Why Stopped: study changed waiting renew
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Lu, Director, Fundus Disease Center of Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2016HM-MF
Record Dates: First submitted 2016-09-04; First posted 2016-09-26 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: High Myopia
Keywords: high myopia; myopia foveoschisis; macular buckling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- MF-MB: Consecutive participants with high myopic foveoschisis are scheduled to macular buckling (MB) surgery.
  Interventions: Procedure: macular buckling surgery

INTERVENTIONS:
Procedure: macular buckling surgery — Participants with high myopia foveoschisis are scheduled to macular buckling (MB) surgery.

SUMMARY:
Macular foveoschisis (MF) is a common complication of pathological myopia, which is characterized by choroid-retinal degeneration and vision impairment. Although pars plana vitrectomy (PPV) is the primary method for MF treatment, there is still a large proportion of recurrent MF due to the extremely long global axial length and posterior staphyloma. Macular buckling (MB) surgery aims at counteracting the traction exerted by the posterior staphyloma, and has been proven an effective method for treating MF. Optical Coherence Tomography (OCT) is widely used for the structural analysis of MF. Multifocol electroretinogram (mfERG) is an objective examination for visual evaluation. To our knowledge, there is a lack of data on the comprehensive visual function evaluations of MF patients associated with OCT findings. Our clinical trial aims to provide the structural and functional relationship in MF patients undergoing MB surgery, and find out potential factors to determine the visual prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. axial length ≥ 26.5 mm or refractive error (spherical equivalent) ≥ 8.0 diopter;
2. macular foveoschisis that requires surgical intervention.

Exclusion Criteria:

1. ocular trauma or surgery history;
2. glaucoma, diabetic retinopathy;
3. intraocular active hemorrhage or inflammation;
4. unable to coordinate the OCT, mfERG, or other ophthalmological examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive participants with high myopia associated macular foveoschsis, who scheduled for surgery at Zhongshan Ophthalmic Center, Sun Yat-sen University.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-12 (Estimated); Study Completion 2021-09-18 (Estimated)

PRIMARY OUTCOMES:
change from baseline OCT at 6 months | 6 month postoperatively
change from multifocal ERG at 6 months | 6 month postoperatively

SECONDARY OUTCOMES:
change from Best-corrected visual acuity (BCVA) at 6 months | 6 month postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided